CLINICAL TRIAL: NCT02566395
Title: A Two Step Approach to Allogeneic Hematopoietic Stem Cell Transplantation From HLA Partially-Matched Related Donors for Patients With Hematologic Malignancies
Brief Title: Stem Cell Transplantation From HLA Partially-Matched Related Donors for Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: New York Blood Center (Other)
Responsible Party: Principal Investigator, Joel Brochstein, Associate Chief for Cellular Therapy, CCMC, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-551
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Chronic Myelogenous Leukemia; Non-Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Stem Cell Transplantation; Haploidentical Donors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Radiation; Whole-Body Irradiation; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Haploidentical Stem Cell Transplantation (Experimental): Subjects will receive pretransplantation conditioning of total-body irradiation (1,200 cGy delivered in 8 fractions over 4 days [Days -9 through -6] and cyclophosphamide (60 mg/kg IV daily x 2 on Days -3 and -2). Donor lymphocyte infusion will occur on day -6; donor CD34+ cells will be infused on Day 0.
  Interventions: Radiation: Radiation; Drug: Cyclophosphamide; Biological: Donor Lymphocyte Infusion (DLI); Biological: Haploidentical Stem Cell Transplantation

INTERVENTIONS:
Radiation: Radiation — 1,200 cGy, delivered in 8 fractions of 150 cGy bid x 4 days
  Other Names: Total Body Irradiation
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg IV daily x 2 consecutive days
  Other Names: Cytoxan
Biological: Donor Lymphocyte Infusion (DLI) — DLI containing 1 x 10E8/kg donor T-cells
Biological: Haploidentical Stem Cell Transplantation — 2-10 x 10E6/kg donor CD34+ selected cells

SUMMARY:
This clinical pilot trial is intended to evaluate the feasibility, efficacy and safety of hematopoietic stem cell transplantation (HSCT) from Human Leukocyte Antigen (HLA)-mismatched related donors for children and young adults with hematologic malignancies who lack a suitably matched related or unrelated donor. The methodology will be one that has been successfully utilized in adult patients at Thomas Jefferson University.

DETAILED DESCRIPTION:
Allogeneic HSCT is a potentially curative therapy for a number of malignancies. A barrier to the institution of this potentially curative strategy in hematologic malignancies is the availability of donors. Only 30% of patients in North America or Europe who may benefit from allogeneic HSCT will have an available HLA matched sibling donor. The ability to find a matched sibling donor is proportional to the number of children in the family. Because of the decreasing size of nuclear families, it is becoming less likely for patients to have an HLA identical matched sibling. Registries can provide a matched unrelated allogeneic stem cell graft for an additional 30% of patients. However this is not an option for patients who do not have a match in the registry, or whose disease status precludes them from waiting to identify an appropriate unrelated donor. The ability of finding a well matched unrelated donor is even more limited for segments of the population with mixed race ancestry as well as for African Americans who, because of a higher degree of HLA diversity, will be unlikely to find an unrelated donor who matches their HLA type.

In these settings it is easier and faster to identify a partially HLA-matched (or haploidentical) family member as a stem cell donor. The use of haploidentical donors broadens the application of HSCT because it is not as limited by family size or racial/ethnic HLA diversity. Because parents and children, as well as siblings can be used as haploidentical donors, this type of transplant enfranchises almost every segment of the population.

Since, in this study, the donor lymphoid and stem cell portions of the graft are collected and administered at different time points during the conditioning regimen, this approach to haploidentical HSCT is referred to as a 2 Step regimen. The approach does not involve ex vivo T cell depletion, but uses cyclophosphamide to tolerize donor lymphocytes within the framework of a myeloablative conditioning regimen. Preliminary experience with this approach in adult patients at Thomas Jefferson University for myeloablative haploidentical HSCT dates back to 2005 with the first trial using myeloablative conditioning formally launched in 2006. That initial trial met its accrual goals and the current trial is one of the successor trials derived from that experience.

The conditioning regimen includes total body irradiation (TBI) (1.5 Gray x 8) and CY (60 mg/kg x 2). Tacrolimus and Mycophenolate Mofetil (MMF) are used as post-transplant immunosuppression in relatively standard fashion.

The novel aspect of the regimen is in the administration of the graft. If one considers that a standard allograft consists of two components, a lymphoid portion and a stem cell portion, what is unique here is the administration of these two portions separately, at different time points during the conditioning regimen rather than together. The lymphoid portion, including a fixed dose of CD3+ cells/kg is administered prior to cyclophosphamide while the hematopoietic stem cell (HSC) portion of the graft is administered after cyclophosphamide has been metabolized and eliminated. Thus, the transplant occurs in 2 steps.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia
* Acue myelogenous leukemia
* Myelodysplastic syndrome
* Non-Hodgkin lymphoma
* Chronic myelogenous leukemia
* Adequate lung, liver, renal, cardiac function
* Performance status >70
* Available related donor who is mismatched at ≥ 2 HLA alleles

Exclusion Criteria:

* Available HLA-identical related donor
* HIV positive
* Active uncontrolled infection
* Pregnancy
* Performance status ≤70

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2022-01-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Hematopoietic engraftment | Day +30 post-transplantation
  Absolute neutrophil count >500/microliter x 3 consecutive days

SECONDARY OUTCOMES:
2-Year disease-free survival | 2 years post-transplantation
  Alive and free of disease at 2 years post-transplantation
Grade II-IV GvHD | Day +100 post-transplantatation
  Proportion of subjects with Grade II-IV acute graft-versus-host disease
Grade III-IV GvHD | Day +100 post-transplantation
  Proportion of subjects with Grade III-IV acute graft-versus-host disease
Relapse rate | 2 years post-transplantation
  Proportion of subjects who have experienced disease relapse by 2 years post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Joel A Brochstein, MD, Principal Investigator — Cohen Children's Medical Center
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

REFERENCES:
- [Background] Grosso D, Gaballa S, Alpdogan O, Carabasi M, Filicko-O'Hara J, Kasner M, Martinez-Outschoorn U, Wagner JL, O'Hara W, Rudolph S, Chervoneva I, Colombe B, Farley PC, Flomenberg P, Pro B, Sharma M, Shi W, Weiss M, Flomenberg N. A two-step approach to myeloablative haploidentical transplantation: low nonrelapse mortality and high survival confirmed in patients with earlier stage disease. Biol Blood Marrow Transplant. 2015 Apr;21(4):646-52. doi: 10.1016/j.bbmt.2014.12.019. Epub 2014 Dec 23. PMID 25542159